CLINICAL TRIAL: NCT01257386
Title: Comparative Efficacy and Safety Study in Patients With Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tillotts Pharma AG (Industry)
Collaborators: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03010301A; 2007L03525 (Other Grant/Funding Number: SFDA_CTA)
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Active Ulcerative Colitis
MeSH Terms: interventions — Mesalamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asacol® (Experimental): Import Mesalazine
  Interventions: Drug: Asacol®
- Mesalazine (Active Comparator): Marketed Mesalazine
  Interventions: Drug: Mesalazine

INTERVENTIONS:
Drug: Asacol® — 400mg tablets
  Other Names: Import Mesalazine
  Arms: Asacol®
Drug: Mesalazine — 400mg tablets
  Other Names: Marketed Mesalazine
  Arms: Mesalazine

SUMMARY:
To demonstrate that import Mesalazine (Asacol®) is non-inferior to the reference drug, marketed Mesalazine, regarding the primary endpoint (reduction of UC-DAI score)in patients with active ulcerative colitis (UC) treated for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ulcerative Colitis (UC) at active phase who are defined to show Ulcerative Colitis-Disease Activitiy Index (UC-DAI) score of 3 or higher but 8 or less, and bloody stool score of 1 or higher

Exclusion Criteria:

* Patients with serious or higher according to diagnostic critera of seriousness and patients with chronic persistent type and with acute serious type in the classification by clinical course

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 251 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Reduction degree of UC-DAI | Week 8

SECONDARY OUTCOMES:
1) Reduction degree of score of each UC-DAI item 2) Remission rate 3) Effective rate | Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Hospital, Shanghai, China

REFERENCES:
- [Derived] Sun J, Yuan Y. Mesalazine Modified-Release Tablet in the Treatment of Ulcerative Colitis in the Active Phase: A Chinese, Multicenter, Single-Blind, Randomized Controlled Study. Adv Ther. 2016 Mar;33(3):400-9. doi: 10.1007/s12325-016-0303-z. Epub 2016 Feb 22. PMID 26898569